CLINICAL TRIAL: NCT06378918
Title: PILO - Comparison of the Effectiveness of the Simple Puncture Compared to the Incision of an Abscess on the PiLOnidal Sinus
Brief Title: Comparison of the Effectiveness of the Simple Puncture Compared to the Incision of an Abscess on the PiLOnidal Sinus
Acronym: PILO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02791-44
Record Dates: First submitted 2024-04-16; First posted 2024-04-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pilonidal Cyst
Keywords: Pilonidal Cyst; abcess; puncture; incision; intergluteal groove
MeSH Terms: conditions — Pilonidal Sinus; Surgical Wound | interventions — Punctures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- puncture/aspiration (Experimental): The puncture is then carried out using a 16 gauge needle. Antibiotic coverage will be offered.
  Interventions: Procedure: puncture
- abscess incision (Active Comparator): The incision is made in the operating room under general or local anesthesia. The intervention is carried out on an outpatient basis but if necessary, short-term hospitalization is carried out. Daily drying is then carried out with nursing care at home until healing.
  Interventions: Procedure: incision of the abscess

INTERVENTIONS:
Procedure: puncture — Local anesthesia is previously carried out with 2-5 cc of 1% lidocaine. The puncture is then carried out using a 16 gauge needle. Antibiotic coverage will be offered. A work stoppage is recommended until the day after the puncture/aspiration but the duration is left to the discretion of the surgeon. A visit is systematically realised 15 days after the puncture/aspiration with a recommendation for earlier consultation in the event of persistence of redness, discharge, pain or onset of fever. If these symptoms recur or persist, it is recommended to make an incision with packing. In the event of fistulization following the puncture, associated with discharge and skin necrosis, local nursing care is recommended. The definitive resection procedure is then planned 4 to 6 weeks after the puncture/aspiration if the evolution is favorable.
  Other Names: aspiration
  Arms: puncture/aspiration
Procedure: incision of the abscess — This is carried out according to the habits of the department: in the operating room under general or local anesthesia or in consultation (or emergencies) under local anesthesia. The procedure is carried out on an outpatient basis but, if necessary, short-term hospitalization is carried out. Daily drying is then carried out with nursing care at home until healing. A work stoppage is recommended for a period of approximately 10 days. A visit is systematically realised 15 days after the incision with a recommendation for earlier consultation in the event of persistence of redness, discharge, pain or onset of fever. If these symptoms recur or persist, it is recommended to make an incision with packing. The definitive resection procedure is then planned 4 to 6 weeks after the initial operation if the evolution is favorable.
  Other Names: gold standard
  Arms: abscess incision

SUMMARY:
Pilonidal disease is a common disease characterized by the presence of abscess in the intergluteal groove. During periods of abscess, current recommendations are to make a simple incision with daily wicking of the abscess. Direct excision at this time is not recommended because there is a risk of incomplete excision. The principle of directed healing after incision of the abscess results in an average dressing period of 21 days. A definitive resection is recommended after 4 to 6 weeks, when healing has been achieved, in order to limit the risk of infectious recurrence.

An alternative has recently been proposed, consisting of a puncture of the abscess, aimed at emptying it under antibiotic coverage. The major advantage of this treatment is that patients no longer need general anesthesia to flatten the abscess. Although this technique is promising, it is currently not the subject of any published or ongoing randomized controlled study registered on Clinicaltrials.gov.

The research hypothesis is that the two techniques have the same results in terms of recurrence before definitive surgical treatment but that drainage puncture would imply a faster healing time, a lower cost of treatment, a quality of superior support, reduced support time and reduced work stoppage.

DETAILED DESCRIPTION:
This is a single-center, prospective, open-label, randomized study. Patients are screened and included during the emergency room consultation or a scheduled consultation. After verification of the selection criteria and provision of clear, fair and appropriate information, patients are offered to participate in the study. If they accept, consent is signed and randomization is carried out.

The procedure under study is puncture/aspiration. Local anesthesia is previously carried out with 2-5 cc of 1% lidocaine. The puncture is then carried out using a 16 gauge needle. Antibiotic coverage will be offered. A work stoppage is recommended until the day after the puncture/aspiration but the duration is left to the discretion of the surgeon. The patient is systematically reviewed 15 days after the puncture/aspiration with a recommendation for earlier consultation in the event of persistence of redness, discharge, pain or onset of fever. If these symptoms recur or persist, it is recommended to make an incision with packing. In the event of fistulization following the puncture, associated with discharge and skin necrosis, local nursing care is recommended. The definitive resection procedure is then planned 4 to 6 weeks after the puncture/aspiration if the evolution is favorable.

The gold standard procedure is incision of the abscess. This is carried out according to the habits of the department: in the operating room under general or local anesthesia or in consultation (or emergencies) under local anesthesia. The procedure is carried out on an outpatient basis but, if necessary, short-term hospitalization is carried out. Daily wicking is then carried out with nursing care at home until healing. A work stoppage is recommended for a period of approximately 10 days. The patient is systematically reviewed at 15 days with a recommendation for earlier consultation in the event of persistence of redness, discharge, pain or onset of fever. If these symptoms recur or persist, it is recommended to make an incision with packing. The definitive resection procedure is then planned 4 to 6 weeks after the initial operation if the evolution is favorable.

The definitive resection procedure is carried out after the flattening of the abscess has healed. It is recommended to perform resection without closure with nursing-care healing at home with daily packings for 15 days. After the 15-day visit, changing the dressings by wicking is recommended daily until healing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a pilonidal sinus abscess
* Surgical indication for flattening the abscess
* Recurrent or de novo abscess
* Signature of consent to participate in the study

Exclusion Criteria:

* Antibiotic therapy initiated before the emergency room consultation or before the scheduled consultation
* Skin necrosis
* Immunosuppression (drug-related or pathological) or diabetes
* Spontaneous fistulization
* Patients who do not speak French
* Pregnant and/or breastfeeding women
* Patients without social security coverage
* Person deprived of liberty by judicial or administrative decision
* Person subject to psychiatric care under duress
* Person subject to a legal protection measure
* Person unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
healing time | within 6 weeks before resection
  Compare the duration of wound healing between the puncture-aspiration and Incision groups => The healing time is defined by the time between the abscess flattens and the moment the skin is epidermised. In this case, it involves stopping the use of nursing care and stopping dressings. Healing is checked by the investigator using a photo taken by the patient. The date of healing is then recorded by the patient in the logbook. In the event of a recurrence of the abscess, with the need for an incision following the acute episode, the healing time is added to the duration of the previous episode.

SECONDARY OUTCOMES:
Effectiveness of the 2 procedures | 4 weeks
  Effectiveness of the puncture-aspiration and the reference technique in terms of disappearance of symptoms => Effectiveness defined by the disappearance of symptoms and characterized by the disappearance of the inflammatory triad: pain, heat and redness 4 weeks after the initial intervention. Recurrence of the abscess or acute infection before the scheduled definitive resection is considered a failure to resolve symptoms.
Cost-utility analysis | 1.5 months and 10 months
  Efficiency of puncture-aspiration compared to incision by a cost-utility analysis => The cost-utility analysis consists of evaluating the Differential Cost-Utility Ratio at 1.5 months (corresponding to the management of the acute phase) and at 10 months (corresponding to the overall care) from the health system perspective.
Duration of nursing care | within 6 weeks before resection
  Period between the date of emergency consultation and the date of the last visit of a nurse before the definitive resection => The care may be discontinuous or delayed from the urgent intervention, particularly if the abscess to be flattened secondarily after the initial intervention.
Duration of work stoppage | within 6 weeks before resection
  Time between initial intervention and return to work.
Returning to work | within 6 weeks before resection
  The time between the initial intervention and the day on which the patient feels able to resume their professional activity normally => The day on which the patient feels capable of resuming professional activity may be before the date of resumption of professional activity.
Quality of life by the EQ-5D-5L questionnary | within 10 months
  Score assessed by the EQ-5D-5L questionnary during each visit with the surgeon and at each recurrence of the abscess => The EQ-5D-5L is a paper self-completed version that aim to describe and value health across a wide range of disease areas.
  This questionnary, developped by EuroQol group association, is a descriptive system that comprise 5 Dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and each dimension has 5 response Levels (no problems, slight problems, moderate problems, severe problems, unable to/extreme problems)
Healing after definitive resection | 3 months after definitive resection
  Healing after definitive resection is defined by the absence of need for local care associated with the complete epidermization of the resection area carried out with directed healing, 3 months after the definitive resection.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien VENARA, PHD, Principal Investigator — University Hospital of Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Parades V, Bouchard D, Janier M, Berger A. Pilonidal sinus disease. J Visc Surg. 2013 Sep;150(4):237-47. doi: 10.1016/j.jviscsurg.2013.05.006. Epub 2013 Aug 1. PMID 23911903
- [Background] Segre D, Pozzo M, Perinotti R, Roche B; Italian Society of Colorectal Surgery. The treatment of pilonidal disease: guidelines of the Italian Society of Colorectal Surgery (SICCR). Tech Coloproctol. 2015 Oct;19(10):607-13. doi: 10.1007/s10151-015-1369-3. Epub 2015 Sep 16. PMID 26377583
- [Background] Doll D, Friederichs J, Boulesteix AL, Dusel W, Fend F, Petersen S. Surgery for asymptomatic pilonidal sinus disease. Int J Colorectal Dis. 2008 Sep;23(9):839-44. doi: 10.1007/s00384-008-0476-2. Epub 2008 May 20. PMID 18491116
- [Background] Doll D, Friederichs J, Dettmann H, Boulesteix AL, Duesel W, Petersen S. Time and rate of sinus formation in pilonidal sinus disease. Int J Colorectal Dis. 2008 Apr;23(4):359-64. doi: 10.1007/s00384-007-0389-5. PMID 18043929
- [Background] Fahrni GT, Vuille-Dit-Bille RN, Leu S, Meuli M, Staerkle RF, Fink L, Dincler S, Muff BS. Five-year Follow-up and Recurrence Rates Following Surgery for Acute and Chronic Pilonidal Disease: A Survey of 421 Cases. Wounds. 2016 Jan;28(1):20-6. PMID 26824973
- [Background] Hussain ZI, Aghahoseini A, Alexander D. Converting emergency pilonidal abscess into an elective procedure. Dis Colon Rectum. 2012 Jun;55(6):640-5. doi: 10.1097/DCR.0b013e31824b9527. PMID 22595842
- [Background] Lasithiotakis K, Aghahoseini A, Volanaki D, Peter M, Alexander D. Aspiration for acute pilonidal abscess-a cohort study. J Surg Res. 2018 Mar;223:123-127. doi: 10.1016/j.jss.2017.09.051. Epub 2017 Nov 17. PMID 29433863